CLINICAL TRIAL: NCT01404299
Title: Effects of a Protein-Energy Nutritional Supplementation on the Functional Status of Frail Older Adults With Low Socioeconomic Status: A Community-based Randomized Trial
Brief Title: Effects of a Nutritional Supplementation on the Functional Status of Frail Elders With Low Socioeconomic Status (SES)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangbuk-gu Community Health Center (Other Government)
Responsible Party: Principal Investigator, Dr. Chang-O Kim, Home Visit Doctor, Gangbuk-gu Community Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GCHC_FRAIL
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Frail
Keywords: Frailty,; nutritional supplementation,; functional status
MeSH Terms: conditions — Frailty | interventions — Dietary Supplements; Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supplementary Group (Experimental)
  Interventions: Dietary Supplement: Nutritional Supplementation
- Control Group (No Intervention)
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Nutritional Supplementation — - Providing two 200mL per day of commercial liquid formula cans for 12 weeks (additional 400kal of energy, 25g of protein, 9.4g of essential amino acids (60.2% leucine), 400mL of water, and micronutrients per day)
  Other Names: Greenbia HP (Dr. Jung's Food Co., Ltd., Korea)
  Arms: Supplementary Group
Other: Control — - No intervention, except monthly home visits
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine whether protein-energy nutritional supplementation improves geriatric function in community-dwelling frail older adults of low socioeconomic status.

DETAILED DESCRIPTION:
Chronic undernutrition is a common condition in older people, and is clearly an important component of frailty. However, the effect of protein-energy nutritional supplementation on the functional status of frail older people is controversial. Some investigators suggested that, if nutritional or functional status has deteriorated too far, it could be very difficult for single nutritional supplementation to reverse malnutrition progression or functional decline.

The investigators believe one of the reasons for these ineffective results, especially for the community-dwelling frail elderly, may be due to a lack of regard to the socioeconomic status of the study population. For this reason, the investigators recruited a study sample with low socioeconomic status and evaluated the effect of protein-energy nutritional supplementation on their disability scores and physical performance.

ELIGIBILITY:
Inclusion Criteria:

* Older adults over 65 years of age, registered in the National Home Healthcare Service database
* Require more than 5 seconds to perform 3m walking test (Usual Gait Speed <0.6 m/sec)
* Get less than 24 points on Mini Nutritional Assessment (Mini Nutritional Assessment <24)

Exclusion Criteria:

* Unable to walk or are too functionally deteriorated to receive home health care services
* Who were participating in any kind of exercise program or clinical nutrition program
* who were restricted to a high-protein diet by an internist (i.e., for liver failure or severe renal failure)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Functional Status | 12 weeks
  Physical Functioning (Self-reported disability score which was specially developed to measure geriatric function in the community-dwelling frail elderly of Korea), Short Physical Performance Battery (Objective measurement of functional performance developed at the Established Population for Epidemiologic Studies of the Elderly)

SECONDARY OUTCOMES:
Nutritional Status, Other Functionality Test | 12 weeks
  Dietary Intake Data, Body Weight, Mid-arm Circumference, Hand Grip Strength, Timed-up-and-go Test, Usual gait speed, One Leg Stands, BUN (Serum), Creatinine (Serum)

CONTACTS AND LOCATIONS:
Overall Officials: Chang-O Kim, M.D, MSW, Study Director — Department of District Health Care Service, Gangbuk-gu Community Health Center, Republic of Korea
Locations (1):
- Gangbuk-gu Community Health Center, Seoul, Seoul, South Korea